CLINICAL TRIAL: NCT04145804
Title: Evaluation Of Hybrid Closed Loop (HCL) System On-Boarding Protocol, For Patients With Type 1 Diabetes On Multiple Daily Insulin Injections (MDI) Therapy
Brief Title: Hybrid Closed Loop System for Patients on Multiple Daily Insulin Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Sidra Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-19-296
Record Dates: First submitted 2019-10-20; First posted 2019-10-31 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes
Keywords: Time in range; Hybrid closed loop system; Multiple daily insulin injection
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Medtronic Minimed 670G insulin pump — It is an insulin pump to deliver insulin to the patient and associated with a sensor to monitor the glucose levels of the patient. The new feature in this device is the automode algorithm which regulates insulin delivery to the patient automatically to keep glucose levels within target.

SUMMARY:
The objective of this study is to assess structured group education onboarding protocol of the 670 G Hybrid Closed Loop (HCL) systems in achieving glucose control of patients on Multiple Daily Insulin Injections (MDI).

DETAILED DESCRIPTION:
Goal

The objective of this study is to assess structured group education onboarding protocol of the 670 G Hybrid Closed Loop systems in achieving glucose control of patients on MDI.

Methods

This study is a single-arm, single-center, clinical investigation in subjects with type 1 diabetes on HCL insulin pump (Minimed 670G) in a period of 3 months. A total of 40 subjects (age 18-65) will be enrolled in order to reach 34 subjects who will complete the HCL study. The investigators will start the clinical process for initiating an insulin pump, which is typically done with pre-pump classes. HbA1c, derived from Continuous Glucose Monitoring (CGM) will be performed at baseline and at the end of the 3-month study period. The following parameters will be analyzed" % patients achieving glucose readings Time in Range (TIR) > 67% in (70-180 mg/dl); % patients achieving <3% Time below Range ( <70 mg/dl) and % patients achieving both TIR > 67% and <3% Time below Range.Collection of demographics and medical history, data for diabetes devices (eg meters, sensors, pumps) and brief clinical physical exam including vital signs and skin assessment will be obtained via Hospital Electronic Medical File (Cerner Millennium) and will be kept as electronic data on a separate research server.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. HbA1c < 12.5%
3. Age18-65 years at the initiation of the 670G system
4. Multiple Daily Injections (Basal Bolus therapy) with Total daily insulin use of great than 8.0 units per day over a 1 week period
5. Willing and able (access to internet from home) to download information into the Medtronic CareLink software
6. Clinically planning to and be able to start the Medtronic 670G HCL system
7. History of 3 clinic visits in the last year
8. With history of cardiovascular event 1 year or more from the time of screening, must have clearance from a cardiologist.

Exclusion Criteria:

1. Diabetic Ketoacidosis in the 6 months prior to screening visit
2. Type 2 diabetes
3. Hyperthyroidism at time of screening
4. Using Pramlintide, Dipeptidyl peptidase 4 (DPP-4) inhibitor, Glucagon-like peptide-1 (GLP-1) agonists, metformin, sodium-glucose transport protein 2 (SGLT2) inhibitors at time of screening.
5. Has taken any oral, injectable, or intravenous (IV) steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The achievable percentage of time in range (TIR) 70 - 180 mg/dL for the whole study population after 3 months. | 3 months
  The achievable Time in Range (TIR) in the first 3 months of MiniMed 670G following onboarding of MDI to HCL by the protocol in a real-life setting.

SECONDARY OUTCOMES:
percentage of patients achieving TIR > 67% in Time in Range (70-180 mg/dl) | 3 months
percentage of patients achieving TIR <3% Time below Range ( <70 mg/dl) | 3 months
percentage of patients achieving both TIR > 67% and <3% Time below Range | 3 months
Change in HBA1C from baseline | 3 months
  Change in HbA1c levels from previous treatment (multiple daily injections) compared to Minimed 670G treatment
Change in sensor glucose values from baseline | 3 months
  Change in sensor glucose values from previous treatment (multiple daily injections) compared to Minimed 670G treatment
Percentage of time above Range (>180 mg/dl) for the whole study population | 3 months
  Percentage of glucose values more than 180 mg/dl on Minimed 670G
Number of severe hypoglycemia episodes | 3 months
Number of Diabetic Ketoacidosis episodes | 3 months
Total daily insulin dose | 3 months
Percentage of time spend in Auto Mode | 3 months
  Percentage of time in Auto Mode, where Minimed 670G automatic adjusts the basal insulin dose according glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Dabia Al Mohanadi, MD, FRCPC, Principal Investigator — Hamad Medical Corporation; Goran Petrovski, MD, PhD, Principal Investigator — Sidra Medicine
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No